CLINICAL TRIAL: NCT02944591
Title: Evaluation of COPD Co-Pilot
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: HGE Health Care Solutions, LLC (Industry)
Collaborators: PneumRx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CPV2-2016-S2
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: COPD Co-Pilot — The COPD Co-PilotTM is a smartphone application for symptom reporting supported by a Call Center staffed with pulmonary nurses and Health Assistants who are trained to support patients with COPD. The call center staff are employees and subcontractors of the company that makes the COPD Co-PilotTM, HGE. It is located on the Campus of Temple University in Philadelphia Pennsylvania.

SUMMARY:
The purpose of this research study is to investigate the potential benefits of participant use of a smartphone application ("App") called COPD Co-Pilot™. When used by the participant, COPD Co-Pilot™ may provide early detection of worsening COPD symptoms. Early symptom detection may allow the pulmonary providers and nurses to respond with timely medical advice and treatment. The goal for use of COPD Co-Pilot™ is to reduce the frequency and duration of hospitalizations, emergency department visits, and hospital readmissions. The study will also examine the financial impact of the COPD Co-Pilot™ program to determine whether costs of hospital stays, emergency department visits, and hospital readmissions differ when patients are enrolled in COPD Co-Pilot™ than when they are not enrolled. Another purpose of this study is to measure patient satisfaction with use of COPD Co-Pilot™.

DETAILED DESCRIPTION:
During the 6-month observational period, subjects will report respiratory symptoms using COPD Co-Pilot on a daily basis and will receive feedback and clinical recommendations from their health care provider when their symptoms change from their baseline symptoms. Final clinical recommendations, medical advice, diagnoses, and treatment are in the full and sole discretion of the provider.

All subjects will receive current standard of care under the supervision of their health care provider. No experimental drugs, dosages, or treatment protocols will be administered at any stage during this trial.

Subjects will receive monthly calls to determine whether any changes to the subject's medical history, hospitalization history, medications, etc. have occurred so they may be added to the subject's profile.

At approximately 6 months post enrollment, all subjects will have an in person end of study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has read, understood and signed an informed consent form prior to enrollment.
2. Males or females age ≥35 years old
3. Documented diagnosis of moderate to very severe COPD (GOLD Level II-IV)
4. Must be able to read and understand English and consent for themselves
5. Subject is willing and able to use an iPad mini device.

Exclusion Criteria:

1. Subject has had an acute exacerbation of COPD that required hospitalization or ER visit or treatment with systemic steroids and/or antibiotics during the 28 days prior to enrollment.

   • Subjects who had a COPD exacerbation within 28 days prior to Visit 1 can be rescreened once. Rescreening can occur no earlier than 28 days from the last dose of systemic steroids and/or antibiotics and/or hospitalization, whichever is later
2. Subject has a COPD exacerbation or respiratory illness during the Run-In period that in the judgment of the investigator requires medical intervention (e.g., treatment with systemic steroids and/or antibiotics and/or hospitalization).

   • Subjects who had a COPD exacerbation or infection during the Run-In period can be rescreened once. Rescreening can occur no earlier than 28 days from the last dose of systemic steroid and/or antibiotics and/or hospitalization, whichever is later.
3. Subject is suffering from terminal illness expected to adversely affect survival in the next 12 months
4. Subject has a history of non-compliance with medical therapies
5. Subject has a cognitive impairment (determined by physician) that will make it hard to follow instructions regarding device usage
6. Subject is currently known to suffer from or have a history of significant substance abuse within the last 2 years
7. Subject has any condition that in the opinion of the provider may adversely affect their participation
8. Subject is residing in hospice care, Skilled Nursing Facilities or Long Term Acute Care facilities
9. Subject has a planned procedures at time of enrollment that will occur within timeframe of study that will require hospitalization or otherwise adversely affect their ability to participate
10. Subject may, in the opinion of the provider, be non-compliant with study schedules or procedures
11. Subject has no cellular coverage at their primary residence
12. Subject plans to travel to a location with no cellular coverage for a significant period (>1 week) during their program participation

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects shall be recruited from the pool of patients at the investigative site that have been diagnosed with moderate to severe COPD.
  The study is planned to enroll 100 subjects. The study will be conducted at one investigative site in the United States, the University of Alabama at Birmingham. Recruitment will stop when 100 subjects are enrolled. There will be no replacement for dropouts. Recruitment is planned to last approximately 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-10; Primary Completion 2018-04-05 (Estimated); Study Completion 2018-04-05 (Estimated)

PRIMARY OUTCOMES:
Patient Adoption | 6 months
  Percentage of potential daily symptom reports completed by patients

SECONDARY OUTCOMES:
Patient Satisfaction | 6 months
  patient satisfaction questionnaire
Inpatient Admissions | 6 months
  admission records for period prior to study and during study
Emergency department visits | 6 months
  emergency department records for period prior to study and during study
Clinic visits | 6 months
  clinic visits for period prior to study and during study
Patient reported respiratory symptoms | 6 months
  Daily values for breathlessness, sputum quantity, sputum color, sputum consistency, peak flow, temperature over 100 F, cough, wheeze, sore throat, and nasal congestion.
Symptom change detected | 6 months
  Change index (a numeric value) and the categorical level of change that corresponds to the patient's reported symptoms when compared to their baseline. This is recorded for each daily symptom report submitted after completion of the run-in period.
Episode duration | 6 months
  the date when a mild, moderate or significant level of change is first detected for a patient through the date immediately followed by seven consecutive days in which a level of "no change" (i.e. return to baseline) is detected. The total number of days in this period, symptoms reported during this period, and clinical responses communicated to the patient (including any treatments or changes) will be reported for analysis.
Time to clinical responses | 6 months
  Time elapsed between the patient's check-in and the time the response was acknowledged by the patient.
Hospitalization history | 6 months
  hospitalization history reported to Health Assistants by patients during scheduled monthly phone calls. This will be reconciled with admissions data from the site and may include utilization at other institutions.
Medications | 6 months
  list of medications and changes entered by site coordinator, provider, or reported by subjects to Health Assistants during scheduled monthly phone calls.
Patient profile information | 6 months
  This will include, among other variables, medical history, smoking history, spirometry results, oxygen use, and diagnoses of co-morbidities. For a full list of profile data, please see the appendix.
Medication compliance | 6 months
  compliance with newly prescribed treatments as reported by patients during follow up phone calls.
Length of stay | 6 months
  total number of inpatient days per admission will be reported for analyses. These records will include date of admission, date of discharge, patient name and medical record number, patient date of birth (DOB), location, length of stay, attending physician, admission diagnosis and diagnosis at discharge. Reported for period prior to study and during study period
Readmissions | 6 months
  The number of inpatient admissions that occur within 30, 60, and 90 days of discharge from a prior admission will be reported for analyses. These records will include date of admission, date of discharge, patient name and medical record number, patient DOB, location, length of stay, attending physician, admission diagnosis, diagnosis at discharge, and associated costs broken down by category. This will be reported for time prior to study and during study period.
Readmission rate | 6 months
  The rate and percent of inpatient admissions that occur within 30, 60, and 90 days of discharge from a prior admission will be reported for analyses. These records will include date of admission, date of discharge, patient name and medical record number, patient DOB, location, length of stay, attending physician, admission diagnosis and diagnosis at discharge. These will be reported for the period prior to the start of the study through the study period.
Source of inpatient admissions and visits to the Emergency Department (ED) | 6 months
  The source (e.g. from home, from accident, from outpatient clinical, at direction of physician, from ED, etc.) of each and every inpatient admission and emergency department visit will be reported for analyses. These will be reported for the period prior to the enrollment through the study period.
Cost of Care | 6 months
  Costs associated with hospitalizations, emergency department visits, clinic visits, and medications
Historic utilization | 6 months
  hospitalizations, emergency department visits, clinic visits in the 6 months prior to enrollment; and hospitalizations, emergency department visits, clinic visits in the same 6 month period during the prior year
Historic costs | 6 months
  costs associated with hospitalizations, emergency department visits, clinic visits in the 6 months prior to enrollment; and costs associated with hospitalizations, emergency department visits, clinic visits in the same 6 month period during the prior year

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Dransfield, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith HS, Criner AJ, Fehrle D, Grabianowski CL, Jacobs MR, Criner GJ. Use of a SmartPhone/Tablet-Based Bidirectional Telemedicine Disease Management Program Facilitates Early Detection and Treatment of COPD Exacerbation Symptoms. Telemed J E Health. 2016 May;22(5):395-9. doi: 10.1089/tmj.2015.0135. Epub 2015 Oct 9. PMID 26451903
- [Background] Cordova FC, Ciccolella D, Grabianowski C, Gaughan J, Brennan K, Goldstein F, Jacobs MR, Criner GJ. A Telemedicine-Based Intervention Reduces the Frequency and Severity of COPD Exacerbation Symptoms: A Randomized, Controlled Trial. Telemed J E Health. 2016 Feb;22(2):114-122. doi: 10.1089/tmj.2015.0035. Epub 2015 Aug 10. PMID 26259074
- [Background] Kim V, Garfield JL, Grabianowski CL, Krahnke JS, Gaughan JP, Jacobs MR, Criner GJ. The effect of chronic sputum production on respiratory symptoms in severe COPD. COPD. 2011 Apr;8(2):114-20. doi: 10.3109/15412555.2011.558546. PMID 21495839
- [Background] So JY, Lastra AC, Zhao H, Marchetti N, Criner GJ. Daily Peak Expiratory Flow Rate and Disease Instability in Chronic Obstructive Pulmonary Disease. Chronic Obstr Pulm Dis. 2015 Nov 11;3(1):398-405. doi: 10.15326/jcopdf.3.1.2015.0142. PMID 28848862
- [Background] Remakus, Christopher B., et al.